CLINICAL TRIAL: NCT05935839
Title: Noninvasive Characterization of Tissue Changes in Diabetes in Adults and Children Using Multispectral Optoacoustic Tomography.
Brief Title: Tissue Changes in Diabetes in Adults and Children Using Multispectral Optoacoustic Tomography.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-205-B
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 1; Macroangiopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Ankle Brachial Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adult Patients with diabetes mellitus type 1 (Experimental): * Laboratory-confirmed diagnosis of diabetes mellitus type 1
  * Age 18-99 years
  * Duration of disease at least 5, preferably 10 years with inadequate medication control (HbA1c value > 8.5 mmol/mol)
  Interventions: Device: Multispectral optoacoustic tomography; Diagnostic Test: Ankle Brachial Index; Diagnostic Test: Neuropathy Disability Score
- Pediatric Patients with diabetes mellitus type 1 (Experimental): * Laboratory-confirmed diagnosis of diabetes mellitus type 1
  * Age 6-17 years
  * Duration of disease at least 5, preferably 10 years with inadequate medication control (HbA1c value > 8.5 mmol/mol)
  Interventions: Device: Multispectral optoacoustic tomography; Diagnostic Test: Ankle Brachial Index; Diagnostic Test: Neuropathy Disability Score
- Healthy volunteers (Experimental): - Age 18-99 years
  Interventions: Device: Multispectral optoacoustic tomography; Diagnostic Test: Ankle Brachial Index; Diagnostic Test: Neuropathy Disability Score

INTERVENTIONS:
Device: Multispectral optoacoustic tomography — Molecular Imaging of tissue changes using MSOT in macroangiopathy in diabetes. Dual imaging before and after physical stress.
Diagnostic Test: Ankle Brachial Index — Dual measurement of ABI index before and after physical exercise.
Diagnostic Test: Neuropathy Disability Score — Single measurement of the NSS

SUMMARY:
In this study, blood flow and tissue changes in adult and pediatric patients with diabetes mellitus will be characterized by MSOT and compared with existing methods (ABI testing, neurological testing) (method comparison). The aim is to quantify changes and to possibly allow early detection of concomitant diseases. This could, similar to peripheral arterial occlusive disease, lead to a new possibility of non-invasive assessment of disease progression in the future.

DETAILED DESCRIPTION:
After informing the patients and parents/guardians and checking the inclusion and exclusion criteria, the clinical data of the ill subjects are recorded and the HbA1c is measured in the laboratory as part of the routine recording. The blood collection is part of the routine diagnostics on presentation in the outpatient clinic and is performed separately from the study.

Subsequently, imaging by MSOT is performed in all study participants. This is performed on both sides of the lower leg over the triceps surae muscle. The examination is analogous to sonography over the corresponding skin layers without further invasive procedures. The anatomical region can be localized by means of built-in sonography; subsequently, the corresponding optoacoustic signals can be derived over it. This is followed by measurement of the Arm-Brachial-Index. After a short recovery time, the test persons perform a physical stress on the examined lower leg muscles. After renewed ABI measurement, the imaging examination is repeated using MSOT. Finally, the neurological status is assessed using the Neuropathy Disability Score (NSS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes mellitus type 1

   * Laboratory-confirmed diagnosis of diabetes mellitus type 1
   * Age 18-99 years
   * Disease duration of at least 5, preferably 10 years with inadequate medication control (HbA1c value > 8.5 mmol/mol)
   * Written informed consent
2. patients with diabetes mellitus type 1

   * Laboratory-confirmed diagnosis of diabetes mellitus type 1
   * Age 6-17 years
   * Duration of disease at least 5, better 10 years with inadequate medication control (HbA1c value > 8.5 mmol/mol)
   * Written informed consent
3. Healthy subjects

   * Age 18-99 years
   * Written informed consent

Exclusion Criteria:

* Pregnancy
* Nursing mothers
* Unstable patients: Need for continuous cardiopulmonary monitoring (ECG and pulse oximetry).
* Tattoo in the area of the examination
* Subcutaneous fat over 3 cm
* Lack of written consent
* Inability to perform sufficient (brief) physical exertion

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Visualization of tissue changes in diabetic patients using MSOT. | 12 months
  Comparison of the quantitative percentage of oxygenated/deoxygenated hemoglobin determined by MSOT in adults and children with diabetes mellitus and an adult healthy control group.